CLINICAL TRIAL: NCT02194582
Title: Molecular and Genetic Analysis of Inherited Kidney Dysfunction
Brief Title: Genetic Causes of FSGS, Nephrotic Syndrome, or Kidney Failure
Acronym: FSGS
Status: Active, not recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Martin R. Pollak, Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2009P000430; 5R01DK054931-18 (NIH)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Focal Segmental Glomerulosclerosis; Nephrotic Syndrome; End Stage Renal Disease; Kidney Failure; Unexplained Proteinuria
Keywords: FSGS; NS; Kidney disease; Kidney failure; Renal disease; nephrotic syndrome; focal segmental glomerulosclerosis; familial kidney disease; minimal change disease; proteinuria
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrotic Syndrome; Kidney Failure, Chronic; Renal Insufficiency; Kidney Diseases; Nephrosis, Lipoid; Proteinuria

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Usually saliva In some cases, a blood sample may be obtained In some cases, a urine sample may be requested
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are trying to learn more about the cause of kidney diseases such as Focal Segmental Glomerulosclerosis (FSGS) and Nephrotic syndrome by studying genetics. The investigators are interested in discovering which genes play a role in causing a predisposition to FSGS/NS. The investigators also want to learn why FSGS/NS can run in families. Participation in our study involves a saliva sample and a urine sample that you can give from home. There is no cost to participate. All information is kept private and confidential. The investigators also like to include healthy volunteers (parents, spouses) if interested/available but of course this is completely optional.

DETAILED DESCRIPTION:
The investigators welcome anyone (with or without a family history) with unexplained, non syndromic FSGS, nephrotic syndrome, or proteinuria to join the study. Participation involves a saliva (or blood if it is preferable) sample and urine sample (if applicable). There is no cost to participate and the study can be done from home in most cases.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with FSGS (focal segmental glomerulosclerosis)
* Subjects with NS (nephrotic syndrome)
* Subjects with unexplained kidney failure (have had a transplant or on dialysis)
* Subjects with unexplained proteinuria
* Family members of a person with FSGS, NS, kidney failure, or unexplained protein in their urine
* Healthy volunteers

Exclusion Criteria:

* Patients whose kidney disease is already explained by another syndrome such as (Branchio Oto Renal Syndrome or Alports syndrome)
* Patients who already know the genetic cause of their kidney disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We are recruiting subjects who have kidney disease, family members of a person with kidney disease, and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 2050 (Estimated)
Dates: Start 1996-06 (Actual); Primary Completion 2035-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
To identify the genetic causes of FSGS, NS, and idiopathic proteinuria/ESRD in patients and families | 2035
  This is an ongoing study for research purposes only.

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Pollak, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States

REFERENCES:
- See also: BIDMC - Pollak Lab Website — https://sites.google.com/site/pollakfsgs/